CLINICAL TRIAL: NCT01262105
Title: Reduction of Airborne Microbes in the Surgical Field During Spine Procedures Using Directed Local Airflow
Brief Title: Device to Reduce Surgery Site Contamination - Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nimbic Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ABS-002
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Surgery
Keywords: CFU; surgery site

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- No device (No Intervention)
- Device deployed (Experimental)
  Interventions: Device: Air Barrier System Device

INTERVENTIONS:
Device: Air Barrier System Device — Device is deployed adjacent to the surgery site and activated so that the filtered air emits over the site.
  Arms: Device deployed

SUMMARY:
The objective of this study is to determine whether the Air Barrier System device reduces airborne colony-forming units (e.g. bacteria) present at a surgery site during spinal procedures.

DETAILED DESCRIPTION:
The Air Barrier System is a device that uses localized clean air flow to shield a surgery site from ambient airborne contamination. This study examines the hypothesis that the Air Barrier System can reduce the presence of airborne colony-forming units at the surgery site during spinal procedures.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for instrumented posterior lumbar interbody fusion

Exclusion Criteria:

* Prior history of infection
* Revision surgery
* Screens positive for MRSA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wimberley, MD, Principal Investigator — Fondren Orthopaedic Group
Locations (1):
- Texas Orthopedic Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Stocks GW, Self SD, Thompson B, Adame XA, O'Connor DP. Predicting bacterial populations based on airborne particulates: a study performed in nonlaminar flow operating rooms during joint arthroplasty surgery. Am J Infect Control. 2010 Apr;38(3):199-204. doi: 10.1016/j.ajic.2009.07.006. Epub 2009 Nov 12. PMID 19913327

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Device | Device Deployed
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Device | Device Deployed | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Surgery Site CFU Density
Description: CFU culture counts for samples taken in surgery.
Time Frame: Ten-minute intervals throughout procedure
Measure: Mean (95% Confidence Interval); unit: CFU/m3
Groups:
- No Device: No device is deployed during surgery
- Device Deployed: The ABS device is employed during surgery.
Arm/Group | No Device | Device Deployed
Number analyzed (Participants) | 13 | 10
CFU/m3 | 3.08 [2.44 to 3.72] | 1.73 [1.03 to 2.43]

ADVERSE EVENTS:
Arm/Group | No Device | Device Deployed
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes